CLINICAL TRIAL: NCT01050543
Title: A Randomized Safety-Assessor Blinded Trial Comparing Sugammadex With Neostigmine in Korean Subjects Scheduled for Surgeries Requiring Moderate Neuromuscular Blockade
Brief Title: Comparison of Sugammadex With Neostigmine as Reversal Agents for Rocuronium at Reappearance of T2 (Study P06101)
Acronym: DANCHEONG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P06101
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental)
  Interventions: Drug: sugammadex
- Neostigmine (Active Comparator)
  Interventions: Drug: neostigmine

INTERVENTIONS:
Drug: sugammadex — sugammadex 2.0 mg/kg, single intravenous bolus dose administered within 10 seconds into a fast flowing venous infusion
  Other Names: SCH 900616; Bridion
  Arms: Sugammadex
Drug: neostigmine — neostigmine 50 mcg/kg (total dose not to exceed 5.0 mg) combined with glycopyrrolate 10 mcg/kg, single intravenous bolus dose administered within 10 seconds into a fast flowing venous infusion
  Other Names: neostigmine methylsulfate
  Arms: Neostigmine

SUMMARY:
This is a randomized, active-controlled, parallel-group, single-dose, multi-site, safety-assessor blinded study comparing sugammadex to neostigmine for reversal of neuromuscular blockade in Korean subjects undergoing elective surgical procedures under general anesthesia that require rocuronium for neuromuscular blockade. Study medication will be administered at reappearance of T2. Time to recovery will be measured from start of study medication administration to recovery of the T4/T1 ratio of 0.9. The primary hypothesis is that the time to recovery of the T4/T1 ratio of 0.9 is shorter with sugammadex than with neostigmine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Class 1 or 2 or 3
* >=18 years of age and of either sex
* scheduled for elective surgical procedure under general anesthesia requiring the use of rocuronium for endotracheal intubation and/or maintenance of neuromuscular blockade in a supine position allowing neuromuscular transmission monitoring and requiring reversal of neuromuscular blockade
* Korean descent born in Korea, never emigrated out of Korea, and have a Korean home address

Exclusion Criteria:

* expected difficult intubation due to anatomic malformations
* expected transfer to intensive care unit after surgery
* neuromuscular disorders affecting neuromuscular blockade
* significant hepatic or renal dysfunction
* require use of pneumatic tourniquet during surgery
* (family) history of malignant hyperthermia
* allergy to cyclodextrins (including sugammadex) or other medication(s) used during general anesthesia; use of toremifene or fusidic acid within 24 hours of study drug administration; contraindication to use of neostigmine or glycopyrrolate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-08-20 (Actual); Study Completion 2010-08-20 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Woo T, Kim KS, Shim YH, Kim MK, Yoon SM, Lim YJ, Yang HS, Phiri P, Chon JY. Sugammadex versus neostigmine reversal of moderate rocuronium-induced neuromuscular blockade in Korean patients. Korean J Anesthesiol. 2013 Dec;65(6):501-7. doi: 10.4097/kjae.2013.65.6.501. Epub 2013 Dec 26. PMID 24427455

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: sugammadex 2 mg/kg
- Neostigmine: neostigmine 50 mcg/kg
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 64 (Includes 4 participants who were randomized but discontinued before Treatment Phase.) | 64 (Includes 4 participants who were randomized but discontinued before Treatment Phase.)
Completed | 60 (Includes 1 participant who started & completed the study but was excluded from Full Analysis Set.) | 60 (Includes 1 participant who started & completed the study but was excluded from Full Analysis Set.)
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Administrative | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (14.0) | 42.6 (14.0) | 42.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Study Drug Administration to Recovery of the T4/T1 Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 & T4 refer to the magnitudes (height) of the 1st & 4th twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade. In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated complete recovery.
Time Frame: From Start of Study Drug Administration to Recovery of the T4/T1 Ratio to 0.9 (estimated from 2 minutes up to ~15 minutes)
Population: Full Analysis Set, defined as all participants who received randomized treatment and had at least one efficacy measurement.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 59 | 59
minutes | 1.77 [1.57 to 2.01] | 14.80 [12.43 to 17.62]
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; To evaluate the efficacy of sugammadex compared to the efficacy of neostigmine, the ratio of the geometric means of time to recovery of the T4/T1 ratio to 0.9 was calculated using a 2-way ANOVA model adjusted for trial site; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [6.8 to 9.6]

ADVERSE EVENTS:
Arm/Group | Sugammadex | Neostigmine
Serious Adverse Events (participants affected / at risk) | 2/60 | 2/60
Other Adverse Events (participants affected / at risk) | 36/60 | 42/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=60) | Neostigmine (N=60)
Post-operative abscess (Infections and infestations) | 1 (1) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=60) | Neostigmine (N=60)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Incision site pain (Injury, poisoning and procedural complications) | 7 (9) | 12 (16)
Procedural hypotension (Injury, poisoning and procedural complications) | 4 (6) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 20 (22) | 18 (19)
Wound complication (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 7 (8) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall have the right to review and comment with respect to publications with regard to the following concerns: proprietary information; accuracy of the information; and to ensure that the presentation is fairly balanced and in compliance with FDA regulations.

The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.